CLINICAL TRIAL: NCT06118268
Title: iTBS to Enhance Social Cognition in People With Psychosis
Acronym: iSCIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Wellcome Trust (Other); Centre for Addiction and Mental Health (Other); University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Anil K. Malhotra, Vice Chair Research, Zucker Hillside Hospital, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-0071
Record Dates: First submitted 2023-10-04; First posted 2023-11-07 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Schizophreniform Disorders; Psychosis Nos/Other
Keywords: TMS; iTBS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active iTBS (Active Comparator)
  Interventions: Device: iTBS (Active)
- Sham iTBS (Sham Comparator)
  Interventions: Device: iTBS (Sham)

INTERVENTIONS:
Device: iTBS (Active) — The present study is a double-blind, randomized clinical trial that will examine if iTBS applied to DMPFC improves social cognitive performance compared to sham stimulation
  DMPFC-iTBS will be administered using the MagPro R30 stimulator equipped with a Cool-B70 coil and Qooler fluid-cooling device (MagVenture, Farum, Denmark), positioned under MRI guidance using the Visor 2.0 system (Advanced Neuro Technologies Enschede, Netherlands).
  Arms: Active iTBS
Device: iTBS (Sham) — DMPFC-iTBS will be administered using the MagPro R30 stimulator equipped with a Cool-B70 coil and Qooler fluid-cooling device (MagVenture, Farum, Denmark), positioned under MRI guidance using the Visor 2.0 system (Advanced Neuro Technologies Enschede, Netherlands).
  Arms: Sham iTBS

SUMMARY:
The goal of this clinical trial is to examine if iTBS applied to the DMPFC improves social cognitive performance compared to sham stimulation in people diagnosed with schizophrenia, schizoaffective disorder, schizophreniform disorder, or psychotic disorder not otherwise specified. The main objectives of this trial are:

* Compare changes in social cognitive performance between the active vs. sham treatment groups
* Compare changes in social cognitive network functional connectivity between the active vs. sham treatment groups

Each participant will receive iTBS (active or sham) five days per week for four consecutive weeks. Functional magnetic resonance imaging (fMRI) scans, clinical assessments, and cognitive tests will be performed at pre-treatment, post-treatment, and 6 months after the completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-39 years.
2. DSM-5 diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, or psychotic disorder not otherwise specified (documented by SCID-5).
3. Prescription of antipsychotic medication for at least 60 days and constant dose for 30 days prior to study entry (either first- or second-generation antipsychotics permitted).
4. Able to participate in the informed consent process and provide voluntary informed consent.

Exclusion Criteria:

1. A history of a DSM-5 substance use disorder (other than cannabis, caffeine, or tobacco) within the past six months; or a positive baseline urine drug screen. Only participants meeting for moderate to severe cannabis use disorder will be excluded.
2. Type 1 diabetes mellitus (i.e., insulin-dependent diabetes mellitus with onset < 35 years of age and/or diabetes mellitus that has been complicated by a prior documented episode of ketoacidosis)
3. Acute or unstable medical illness (e.g., delirium, cancer, uncontrolled diabetes, decompensated cardiac, hepatic, renal or pulmonary disease, stroke, or myocardial infarction), whose pathology or treatment could alter the presentation or treatment of schizophrenia or significantly increase the risk associated with the proposed treatment protocol
4. Neurological disease associated with extrapyramidal signs and symptoms (e.g., Parkinson's disease); epilepsy, if the person has had one or more grand mal seizures in the past 18 months; history or physical signs of stroke; any diagnosis of a Central Nervous System (CNS) disorder
5. Requires a benzodiazepine with a dose equivalent to lorazepam 2 mg/day or higher due to the potential of these medications to limit the efficacy of iTBS
6. Suspected DSM-5 intellectual disability based upon clinical interview and psychosocial history
7. Prior Psychosurgery
8. Presence of MRI contraindications (e.g., pacemakers)
9. Pregnancy
10. TMS treatment in the past three months

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in social cognitive performance | From baseline to 4 weeks
  Measured using the emotion recognition (ER-40) task
Change in social cognitive performance | From baseline to 4 weeks
  Measured using the reading the mind in the eyes (RMET) task
Change in social cognitive performance | From baseline to 4 weeks
  Measured using the test of the awareness of social inference-revised (TASIT-R)

SECONDARY OUTCOMES:
Change in social cognitive network functional connectivity | From baseline to 4 weeks
  Measured using the empathic accuracy fMRI task

CONTACTS AND LOCATIONS:
Locations (1):
- Zucker Hillside Hospital, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: No